CLINICAL TRIAL: NCT07298213
Title: Pilot Test of Su Corazon Su Vida Among Mexican Origin Adults With MASLD
Brief Title: Corazones Unidos Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006222
Record Dates: First submitted 2025-12-11; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-06

CONDITIONS: CVD - Cardiovascular Disease; MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corazones Unidos (Experimental): "Corazones Unidos" will be delivered over 12 weekly in-person 60-minute sessions to dyads (consisting on both, intervention and social network participants) in community-based settings.
  Interventions: Behavioral: Your Heart, Your Health
- Su Corazon, Su Vida (Active Comparator): "Su Corazón, Su Vida" group will receive the standard 12-week evidence-based curriculum as a group in a community setting; however, with no peer support provided.
  Interventions: Behavioral: Your Heart, Your Health

INTERVENTIONS:
Behavioral: Your Heart, Your Health — Trained CHWs will facilitate educational sessions where participants will learn about heart-healthy behaviors, heart attack symptoms, heart-healthy eating for Hispanic families, and risk factors for both CVD and MASLD. Participants will also be taught behavioral change techniques including goal setting, problem solving, and relapse prevention. Specifically, participants will be asked to collaborate in selecting specific lifestyle goals and to develop shared strategies for improving adherence to their goals, overcoming barriers, and providing support to address potential relapses. Curriculum content will be supplemented by a variety of approaches designed to motivate behavior change including videos, role play, and low-literacy culturally appropriate brochures published by NHLBI.

SUMMARY:
CVD is the leading cause of death among individuals with MASLD, a risk factor for liver cancer. In Southern Arizona, CVD and cancer (including liver and gastric cancer) are among the leading causes of death for Mexican-origin adults.1 Given Mexican-origin adults' disproportionate burden of CVD-related mortality37 and higher rates of MASLD compared to other ethnic/racial groups; we urgently need to develop contextually tailored strategies for management of CVD risk factors and outcomes. Thus, the purpose of this study is to examine the acceptability and feasibility of a community health worker (CHW)-led intervention aimed to increase cardiovascular risk awareness and promote lifestyle modifications among Mexican-origin adults with Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) in the Southern Arizona region. The proposed project has the potential to improve health outcomes for this vulnerable population and contribute to the ACS-CHERC's overarching goal of improving health equity for Hispanic communities and family caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Eligible intervention participants must (1) be Mexican-origin/Mexican decent, (2) be ≥ 18 years old, (3) have a confirmed MASLD diagnosis (CAP score of ≥ 248 dB/m); (4) have an adult member of their social network who might be interested in participating in the study and who lives within 25 miles of the participant's residence; (5) be able to provide informed consent; and (6) be able to speak, read, and write in English and/or Spanish. Eligible social support participants must (1) be ≥ 18 years old, (2) be first degree blood relative or spouse/significant other to the intervention participants, (3) be able to provide informed consent; and (4) be able to speak, read, and write in English and/or Spanish.

Exclusion Criteria:

* Exclusion for individuals interested in the intervention component of the study will be excluded if they report (1) ongoing or recent alcohol consumption (≥21 standard drinks on average per week in men and ≥14 standard drinks on average per week in women); (2) previous diagnosis of liver cancer; (3) taking any anti-inflammatory or hepatoxic medication regularly; (4) taking medication for any form of psychiatric disorders; (5) diagnosis of depression; (6) diagnosis of autoimmune disorders; or (7) women who are pregnant or breastfeeding due to hormonal changes. Exclusion for those interested to be part of the study as social network participants will not be considered for participation if they (1) live more than 25 miles of the intervention participant's residence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2026-07-17 (Estimated); Study Completion 2026-07-17 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Health | Baseline, 12 weeks, and 24 weeks
  A composite score modeled after the American Heart Association Life's Essential Eight will be computed. Independent scores for diet, physical activity, nicotine exposure, sleep health, body mass index, blood lipids, blood glucose, and blood pressure will be calculated and then transformed into a graded score ranging from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Locations (1):
- UA Collaboratory for Metabolic Disease Prevention & Treatment, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No